CLINICAL TRIAL: NCT05186090
Title: Active Gains in Brain Using Exercise During Aging: AGUEDA Trial
Brief Title: Active Gains in Brain Using Exercise During Aging
Acronym: AGUEDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Instituto Mixto Universitario Deporte y Salud (iMUDS) (Unknown); Centro de Investigación Mente, Cerebro y Comportamiento (CIMCYC) (Unknown); University Hospital Virgen de las Nieves (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Irene Esteban-Cornejo, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RTI2018-095284-J-I00
Record Dates: First submitted 2021-10-17; First posted 2022-01-11 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Healthy; Cognitive Function 1, Social
Keywords: brain; cognition; executive function; exercise; brain-gut axis; positron emission tomography; magnetic resonance imaging; aging; preclinical Alzheimer Disease stages
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24-week resistance exercise program (Experimental): Participants will engage in supervised 24-week resistance exercise program with goal of maintaining 180 minutes of exercise per week.
  Interventions: Behavioral: 24-week resistance exercise program
- Wait-list control group (No Intervention): Control group will be asked to maintain their usual lifestyle.

INTERVENTIONS:
Behavioral: 24-week resistance exercise program — This group will perform a 24-week resistance exercise program. Participants will engage in 180 minutes/week of resistance exercise (3 supervised sessions peer week, 60 min/session). The training will consist of a combination of upper and lower body exercises using elastic bands and participants' body weight as the primary resistance. Exercise load and intensity will be based on the number of repetitions (i.e.,10-12 repetitions), resistance of the elastic bands, in ascending order with seven intensities, and also on the exercises' difficulty (i.e., three levels). The prescribed targeted intensity will reach 70-80% of the participants' maximum rating perceived exertion (i.e., 7-8 RPE).The progression (horizontal) will be standardized according to the execution time and RPE, and individualized according to execution speed and band resistance. Heart rate will be monitored in all sessions. Further, intrinsic motivation before and after session and sleep quality will be registered.
  Arms: 24-week resistance exercise program

SUMMARY:
AGUEDA (Active Gains in brain using Exercise During Aging) is a randomized controlled trial designed to examine the effects of a 24-week resistance exercise program on brain health in cognitively normal adults between 65-80 years of age.

DETAILED DESCRIPTION:
Exercise has emerged as the most promising non-pharmacologic intervention for improving brain health in older adults. The main aim of AGUEDA (Active Gains in brain using Exercise During Aging) trial is to examine the effects of a 6-month resistance exercise program on executive function in cognitively normal older adults. The secondary aims are (i) to examine the effects of exercise on central and peripheral brain markers, and (ii) to investigate mediators and moderators of the exercise-derived improvements observed in executive function and brain markers. AGUEDA is a randomized controlled trial in which 90 cognitively normal older adults, aged 65-80 years old, will be randomized into an exercise group (n=45) or a wait-list control group (n=45). Participants assigned to the exercise group will participate in a 24-week resistance exercise program (3 sessions/week, 60 min/session), while the control group will be asked to maintain their usual lifestyle. A comprehensive neuropsychological test battery, amyloid PET scan, cutting-edge MRI scan, DXA scan, physical ﬁtness, physical function and physical activity measures will be used. Blood, saliva and fecal samples will be collected. Mental health and psychosocial variables will be self-reported.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 65 - 80 years.
* Able to speak and read fluent Spanish.
* Living in community during the study.
* Reliable means of transportation.
* Being physical inactive (i.e., not to be participating in the last 6 months in any resistance exercise program, or accumulating less than 600 METS/Week of moderate-vigorous physical activity).
* Classified as cognitively normal according to Stics-m MMSE and MOCA tests.

Exclusion Criteria:

* Ambulatory with pain or regular use of an assisted walking device.
* Medical contraindication for inclusion in an exercise program.
* Neurological condition (Multiple Sclerosis, Parkinson Disease, Dementia) or brain injury (traumatic or stroke).
* Current diagnosis and treatment of a DSM-V Axis I or II disorder including major depression and seeing a psychologist, therapist, or psychiatrist.
* History of major psychiatric illness including schizophrenia, general anxiety disorder or depression (GDS-30>=15).
* Current treatment for congestive heart failure, angina, uncontrolled arrhythmia, deep venous thrombosis or other cardiovascular event.
* Myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac condition in the past year.
* Current or previous treatment for any type of cancer.
* Type I Diabetes or uncontrolled Type II Diabetes defined as Insulin dependent or Hba1C greater than 10.
* Recent treatment for alcohol or substance abuse.
* Presence of metal implants (e.g., pacemaker, stents, joint replacement) that would be MRI ineligible.
* Claustrophobia.
* Color blindness.
* Diagnosis of COVID-19 with hospitalization in intensive care unit.
* Any other consideration that interferes with the study aims and could be a risk to the participant, at the discretion of the researcher.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Change in executive function | Baseline, 3 months and 6 months
  The main outcome is change in executive function from baseline to 6 months. The 3-month measure is used to assess the trajectory of the change. A comprehensive neuropsychological battery will assess several domains of executive function: working memory, cognitive flexibility and inhibitory control.

SECONDARY OUTCOMES:
Change in brain amyloid beta | Baseline and 6 months
  PET (positron emission tomography) scan using the tracer Neuraceq (Florbetaben F18) will measure levels of the protein amyloid beta in the brain.
Change in brain morphology | Baseline and 6 months
  MRI (magnetic resonance imaging) will measure brain morphology including volume, area, cortical thickness and shapes by a T1-weighted MPRAGE structural sequence.
Change in hippocampal brain morphology | Baseline and 6 months
  MRI (magnetic resonance imaging) will measure hippocampal morphology including volume, area, cortical thickness, shapes by a high resolution hippocampus sequence.
Change in white matter structure | Baseline and 6 months
  MRI (magnetic resonance imaging) will measure white matter structure and lesions by diffusion weighted acquisition sequence.
Change in brain function | Baseline and 6 months
  MRI (magnetic resonance imaging) will measure brain function including both resting state and n-back working memory task-evoked patterns. Measures of brain activity and brain connectivity will be calculated.
Change in cerebral blood flow | Baseline and 6 months
  MRI (magnetic resonance imaging) will measure cerebral blood flow by Pseudo-Continuous Arterial Spin Labeling (pCASL) sequence.
Change in peripheral amyloid beta | Baseline and 6 months
  Saliva and blood samples will be used to determine peripheral amyloid beta
Change in other peripheral neurology biomarkers | Baseline and 6 months
  Saliva and blood samples will be used to determine peripheral neurology biomarkers including brain-derived neurotrophic factor (BDNF), vascular endothelial growth factor (VEGF) and cathepsin B (CTSB).
Change in memory performance | Baseline and 6 months
  Visuospatial memory will be assessed by the Rey-Osterreith figure (ROF) test, verbal memory by the Rey Auditory Verbal Learning Test (RAVLT) and confrontational word memory by the boston Naming Test (short version, BNT).
Change in fluid and crystallized intelligence | Baseline and 6 months
  Intelligence will be assessed by the Wechsler Adult Intelligence Scale (WAIS-IV). 3 subtests for crystallized intelligence (Similarities, Vocabulary, information) and 3 subtests for fluid intelligence (Block Design, Matrix Reasoning, Visual Puzzles).
Change in general cognition | Baseline and 6 months
  General cognition will be assessed by the Telephone Interview for Cognitive Status (STICS-m), the Mini mental state examination (MMSE) and the Montreal Cognitive Assessment (MOCA. vocabulary/language and subjective and objective cognitive decline will be assessed by paper-based tests.
Change in other cognitive outcomes | Baseline and 6 months
  Vocabulary/language, and subjective and objective cognitive decline will be assessed by paper-based tests.

OTHER OUTCOMES:
Changes in muscular strength | Baseline, 3 months (only for field-based tests) and 6 months
  Muscular strength will be assessed by laboratory (i.e. isokinetic test) and field- based (i.e., handgrip and functional tests) tests
Change in physical function | Baseline, 3 months and 6 months
  Senior Fitness Test and Short Physical Performance Battery will assess overall physical functioning and z-scores will be calculated.
Change in gait speed and variability | Baseline and 6 months
  Gait analysis will be assessed by the OptoGait System
Change in cardiorespiratory fitness | Baseline and 6 months
  Cardiorespiratory fitness will be assessed by 2 field-based tests ( i.e., 6-min walking test and 2-km walking test)
Change in mental health outcomes, specifically psychological ill-being | Baseline and 6 months
  A battery of questionnaire will assess psychological ill-being (i.e. depression, anxiety, stress or negative affect).
Change in mental health outcomes, specifically psychological well-being. | Baseline and 6 months
  A battery of questionnaire will assess psychological well-being (i.e. self-esteem, self-concept, self-efficacy, self-image, positive affect, optimism, happiness and satisfaction with life).
Change in quality of life | Baseline and 6 months
  This will be self-reported using the Health Survey Short Form (SF-36).
Change in 24-hours movement behaviors | Baseline and 3 months
  Physical activity at different intensities (average min/day), sedentary time (average min/day) and sleep (average min/day) will be measured using Actigraph GT3X + accelerometers
Change in sedentary behaviors | Baseline and 6 months
  Type of sedentary behaviors will be self-reported by questionnaire.
Change in diet behaviors | Baseline and 6 months
  This will be self-reported using the food-frequency questionnaire (FFQ) and the PREDIMED-14 questionnaire.
Change in body composition | Baseline and 6 months
  Body composition [i.e., lean mass (kg), fat mass (kg), and bone mineral content and density (z-score)] will be assessed using a dual-energy x-ray absorptiometer (DXA). Full- body, bilateral hips and lumbar spine scans will be acquired.
Change in neck adipose tissue | Baseline and 6 months
  Neck adipose tissue will be assessed by MRI
Change in blood pressure | Baseline and 6 months
  Systolic and diastolic blood pressure will be assessed by a blood pressure monitor
Change in peripheral inflammatory and cardiovascular biomarkers | Baseline and 6 months
  Saliva and blood samples will be used to determine peripheral biomarkers including tumor necrosis factor-alpha (TNF-alpha), interleukin-1 beta (IL-1beta), glucose, insulin, HDL and LDL cholesterol
Change in epigenetics and gene expression | Baseline and 6 months
  Blood samples will be stored for genetic analyses, including APOE and BDNF genotypes
Change in oral and gut microbiota | Baseline and 6 months
  Saliva and fecal samples will be used to determine oral and gut microbiota including the most representative phyla (i.e., firmicutes, bacteroidetes, and proteobacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Esteban-Cornejo, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solis-Urra P, Molina-Hidalgo C, Garcia-Rivero Y, Costa-Rodriguez C, Mora-Gonzalez J, Fernandez-Gamez B, Olvera-Rojas M, Coca-Pulido A, Toval A, Bellon D, Sclafani A, Martin-Fuentes I, Trivino-Ibanez EM, de Teresa C, Huang H, Grove G, Hillman CH, Kramer AF, Catena A, Ortega FB, Gomez-Rio M, Erickson KI, Esteban-Cornejo I. Active Gains in brain Using Exercise During Aging (AGUEDA): protocol for a randomized controlled trial. Front Hum Neurosci. 2023 May 22;17:1168549. doi: 10.3389/fnhum.2023.1168549. eCollection 2023. PMID 37284481
- [Background] Fernandez-Gamez B, Solis-Urra P, Olvera-Rojas M, Molina-Hidalgo C, Fernandez-Ortega J, Lara CP, Coca-Pulido A, Bellon D, Sclafani A, Mora-Gonzalez J, Toval A, Martin-Fuentes I, Bakker EA, Lozano RM, Navarrete S, Jimenez-Pavon D, Liu-Ambrose T, Erickson KI, Ortega FB, Esteban-Cornejo I. Resistance Exercise Program in Cognitively Normal Older Adults: CERT-Based Exercise Protocol of the AGUEDA Randomized Controlled Trial. J Nutr Health Aging. 2023;27(10):885-893. doi: 10.1007/s12603-023-1982-1. PMID 37960912
- [Background] Solis-Urra P, Rodriguez-Ayllon M, Alvarez-Ortega M, Molina-Hidalgo C, Molina-Garcia P, Arroyo-Avila C, Garcia-Hermoso A, Collins AM, Jain S, Gispert JD, Liu-Ambrose T, Ortega FB, Erickson KI, Esteban-Cornejo I. Physical Performance and Amyloid-beta in Humans: A Systematic Review and Meta-Analysis of Observational Studies. J Alzheimers Dis. 2023;96(4):1427-1439. doi: 10.3233/JAD-230586. PMID 38007656
- [Background] Rodriguez-Ayllon M, Solis-Urra P, Arroyo-Avila C, Alvarez-Ortega M, Molina-Garcia P, Molina-Hidalgo C, Gomez-Rio M, Brown B, Erickson KI, Esteban-Cornejo I. Physical activity and amyloid beta in middle-aged and older adults: A systematic review and meta-analysis. J Sport Health Sci. 2024 Mar;13(2):133-144. doi: 10.1016/j.jshs.2023.08.001. Epub 2023 Aug 7. PMID 37558161
- [Derived] Fernandez-Gamez B, Solis-Urra P, Coca-Pulido A, Molina-Hidalgo C, Olvera-Rojas M, Bakker EA, Bellon D, Sclafani A, Mora-Gonzalez J, Fernandez-Ortega J, Sanchez-Aranda L, Martin-Fuentes I, Toval A, Sanchez-Martinez J, Wan L, Gomez-Rio M, Liu-Ambrose T, Erickson KI, Ortega FB, Esteban-Cornejo I. Effect of a 24-week resistance exercise intervention on cognitive function in cognitively normal older adults: The AGUEDA randomized controlled trial. Alzheimers Dement. 2026 Jan;22(1):e71019. doi: 10.1002/alz.71019. PMID 41562376
- [Derived] Coca-Pulido A, Solis-Urra P, Fernandez-Gamez B, Olvera-Rojas M, Bellon D, Sclafani A, Toval A, Martin-Fuentes I, Bakker EA, Fernandez-Ortega J, Gomez-Rio M, Hillman CH, Erickson KI, Ortega FB, Mora-Gonzalez J, Esteban-Cornejo I. Fitness, Gray Matter Volume, and Executive Function in Cognitively Normal Older Adults: Cross-Sectional Findings From the AGUEDA Trial. Scand J Med Sci Sports. 2024 Oct;34(10):e14746. doi: 10.1111/sms.14746. PMID 39425451
- See also: AGUEDA website — http://profith.ugr.es/agueda

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT05186090/SAP_000.pdf